Official Title: HIV-Related Stigma Intervention for Malaysian Clinicians NCT number: NCT05597787

Document date: March 29, 2022



#### **PARTICIPANT INFORMATION SHEET**

Study Title: Pilot Test of an Internet-Based HIV Training Program: A Study for

Clinicians. Part 1 Consent

Version No: 2

Version Date: March 29, 2022

We would like to invite you to take part in a research study. Before you decide whether to participate, you need to understand why the research is being done and what it would involve. Please take time to read the following information carefully; talk to others about the study if you wish.

Ask us if there is anything that is not clear or if you would like more information. Take time to decide whether or not you wish to take part.

## 1. What is the purpose of this study?

In the next few months, we will begin pilot testing internet-based HIV training programs for clinicians. Today, we are inviting you to sign up for one of these programs. We are asking you to provide us with some information about yourself. We will use this information to assign you to one of our training programs. We will get back in touch with you with more details about your training program in the next few weeks.

#### 2. Why is this study important?

Many people who are at risk for HIV do not receive HIV tests or prevention counseling in healthcare settings. Additionally, many people who are newly diagnosed with HIV are not linked to HIV care. This study will evaluate whether an internet-based HIV training program can improve clinicians' capacity to provide HIV services to people at risk of or newly diagnosed with HIV.

## 3. What type of study is this?

This is a survey study. We will ask you to answer several questions about yourself.

The next step is an intervention study. You will be randomly assigned to receive one of several types of internet-based HIV training. The training will take place over the period of 9 months, including two one-hour sessions per month. You will be asked to complete several online surveys and an interview to tell us your thoughts about the training.

#### 4. What is the procedure that is being tested?

An internet-based HIV training will be tested in the next step of the study. We will tell you more about the training when we reach back out to you.

## 5. Why have I been invited to participate in this study?

You have been invited to participate in this study because you are 18 or older, a practicing general practitioner or family medicine specialist, and have internet access.

## 6. Who should not participate in the study?

You should not participate in the study if you are unable to join a training session two times per month over lunchtime.

## 7. Can I refuse to take part in the study?

Yes, you can refuse to take part in the study or drop out of the study at any time. If you refuse to take part, your relationships with the University of Malaya and the Ministry of Health will not be affected. There are no penalties for refusing to take part in the study.

#### 8. What will happen to me if I take part?

If you decide to take part in this study, you will be asked to complete a brief survey that includes several questions about yourself and your availability. We will use this information to assign you to a training program, and will contact you within a few weeks with details about your program.

#### 9. How long will I be involved in this study?

It takes about 5 minutes to complete this survey.

#### 10. What are the possible disadvantages and risks?

The main disadvantage of this study is the time it takes to do the survey.

#### 11. What are the possible benefits to me?

You will probably not benefit from completing this survey. If you join a training, you may benefit by receiving some limited specialty training in HIV testing, prevention, and linkage to care.

## 12. Who will have access to my medical records and research data?

Only members of the study team will have access to your research data.

#### 13. Will my records/data be kept confidential?

Yes, we will keep your data confidential. Your name will not be associated with results from this study.

## 14. What will happen if I don't want to carry on with the study?

You can stop participating in the study at any time. You can sign up for a training now and decide that you do not want to participate later.

## 15. What will happen to the results of the research study?

Results of this survey will be used to assign you to a training program.

Results of the intervention study will be analyzed to determine which training program best improves clinicians' capacity to provide HIV services to people at risk of or newly diagnosed with HIV. Results may be shared at scientific meetings and in scientific journals.

## 16. Will I receive compensation for participating in this study?

You will not receive compensation for completing this survey. You will receive incentives and compensation if you participate in a training program.

## 17. Who funds this study?

This study is funded by the National Institute of Mental Health in the United States of America.

# 18. Who should I contact if I have additional questions/problems during the course of the study?

Adeeba Kamarulzaman University of Malaya, Department of Medicine 603-79492050

## 19. Who should I contact if I am unhappy with how the study is being conducted?

Medical Research Ethics Committee University of Malaya Medical Centre Telephone number: 03-7949 3209/2251

BK-MIS-1116-E03